CLINICAL TRIAL: NCT00190034
Title: N-Acetylcysteine Protects Against Acute Renal Insult in Patients With Abnormal Renal Function Undergoing Cardiopulmonary Bypass.
Brief Title: Acetylcysteine Against Acute Renal Insult During Cardiopulmonary Bypass.
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: opposite result
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Synmosa Biopharma Corp. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FEMH-93010; FEMH-93-C-030
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2006-06

CONDITIONS: Cardiovascular Disease; Renal Insufficiency, Acute; Cardiopulmonary Bypass
Keywords: Acetylcysteine; cardiac surgery; cardiopulmonary bypass; acute renal insufficiency
MeSH Terms: conditions — Cardiovascular Diseases; Acute Kidney Injury | interventions — Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine 600mg/tab

SUMMARY:
The purpose of this study is to determine whether N-acetylcysteine is effective in the prophylaxis of post-cardiopulmonary bypass acute renal impairment.

DETAILED DESCRIPTION:
BACKGROUND Reactive oxygen species have been shown to cause contrast-induced nephrotoxicity (CIN). According to previous studies, the N-acetylcysteine has been proved to be advantageous in the avoidance of CIN. We seek to evaluate the efficacy of the antioxidant N-acetylcysteine in limiting the nephrotoxicity after cardiovascular surgery with cardiopulmonary bypass.

METHODS We will prospectively study 60 patients who will receive a cardiovascular surgery with cardiopulmonary bypass. Patients will be randomly assigned to receive either N-acetylcysteine (600 mg orally twice daily for 4 doses) with 0.45% saline intravenously, before and after cardiopulmonary bypass, or placebo with 0.45% saline. Serum creatinine and blood urea nitrogen will be measured before, 48 h and 5 days after the operation procedure.

Expected results Prophylactic oral administration of the antioxidant N-acetylcysteine, along with hydration, will significantly reduce the acute renal damage induced by CPB in patients with chronic renal insufficiency that need cardiovascular procedures.

ELIGIBILITY:
Inclusion Criteria:

* All patients who will received cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

1. Dialyzed patients
2. Acute renal failure
3. Advanced left ventricular systolic dysfunction defined as left ventricular ejection fraction ≦ 35%.
4. Acute chronic obstructive lung disease or asthma exacerbation
5. Allergy to N-acetylcysteine

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-01; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine and blood urea nitrogen: before, 48 h and 5 days after the operation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-jung Li, M.D., Study Chair — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan